CLINICAL TRIAL: NCT06337981
Title: A Phase 2 Multicenter, Randomized, Double-blinded, Placebo-controlled Trial to Evaluate the Efficacy and Safety of AJU-S56 in Patients With Dry Eye Disease
Brief Title: Efficacy and Safety of AJU-S56 in Dry Eye Syndrome Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AJU Pharm Co., Ltd. (Industry)
Collaborators: GL Pharm Tech Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21DE20901
Record Dates: First submitted 2024-03-24; First posted 2024-03-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Dry Eye Syndromes
Keywords: Dry eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test group 1 (Experimental): (AJU-S56 5%) and placebo(Vehicle), 1drop/1times, 3times in a day
  Interventions: Drug: (AJU-S56 5% and placebo)
- Test group 2 (Experimental): (AJU-S56 5%), 1drop/1times, 6times in a day
  Interventions: Drug: AJU-S56 5%
- Comparator group (Placebo Comparator): Placebo(Vehicle), 1drop/1times, 6times in a day
  Interventions: Drug: Placebo(Vehicle)

INTERVENTIONS:
Drug: (AJU-S56 5% and placebo) — (AJU-S56 5%) and placebo(Vehicle), 1drop/1times, 3times in a day
  Other Names: Test 1 group(AJU-S56 5% and placebo, each 1 drop/1time, 3times in a day)
  Arms: Test group 1
Drug: AJU-S56 5% — (AJU-S56 5%), 1drop/1times, 6times in a day
  Other Names: Test 2 group(AJU-S56 5%, 1 drop/1time, 6times in a day)
  Arms: Test group 2
Drug: Placebo(Vehicle) — Placebo(Vehicle), 1drop/1times, 6times in a day
  Other Names: Placebo group(Vehicle, 1 drop/1time, 6times in a day)
  Arms: Comparator group

SUMMARY:
This study is planned to Evaluate the Efficacy and Safety of test drug (AJU-S56) compared to control drug(vehicle) in Patients with Dry Eye Disease.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female who over 19 years old
* Moderate to Severe Dry Eye Disease Patients
* Must meet all criteria listed below at least in one eye or both eyes. TCSS (National eye institute (NEI) scale)≥ 4 Schirmer test(without anesthesia) ≤ 10mm in 5 mins Tear break-up time ≤ 6 secs
* Written informed consent to participate in the trial

Exclusion Criteria:

* Those who have clinically significant eye disease not related to dry eye syndrome
* Those who have medical history with intraocular surgery 12months before screening visit
* Use of corticosteroid, beta blocker and anticholinergic agent within 4 weeks
* Participation in other studies within 4weeks of screening visit

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-11-28 (Actual)

PRIMARY OUTCOMES:
Total corneal staining score (TCSS) | WEEK 4(Visit 4) (*Baseline, Visit 2 is performed in Day 0, Week 0)
  Total corneal staining score (TCSS) ≥4 at baseline (Total Max score : 15, bigger socre means worse outcome)

SECONDARY OUTCOMES:
LGCSS | WEEK 2(Visit 3), 4(Visit 4), 8(Visit 5), 12(Visit 12) (*Baseline, Visit 2 is performed in Day 0, Week 0)
  Lissamine Green Conjunctival Staining Score(Total score : 0~18)
TFBUT | WEEK 2(Visit 3), 4(Visit 4), 8(Visit 5), 12(Visit 12) (*Baseline, Visit 2 is performed in Day 0, Week 0)
  Tear Film Break Up Time

CONTACTS AND LOCATIONS:
Locations (1):
- AJU Pharm Co., Ltd., Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No